CLINICAL TRIAL: NCT03544125
Title: A Pilot Study of Olaparib and Durvalumab in Patients With Metastatic Triple Negative Breast Cancer
Brief Title: Olaparib and Durvalumab in Treating Participants With Metastatic Triple Negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); Prospect Creek Foundation (Unknown)
Responsible Party: Principal Investigator, Zahi Mitri, MD, MS, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00018239; NCI-2018-00819 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00018239 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Estrogen Receptor Negative; HER2/Neu Negative; Progesterone Receptor Negative; Prognostic Stage IV Breast Cancer AJCC v8; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — durvalumab; Immunoglobulin G; Disulfides; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (olaparib, durvalumab) (Experimental): Participants receive olaparib PO twice a day BID for 28 days in the absence of disease progression or unacceptable toxicity. Participants then receive olaparib PO BID on days 1-28 and durvalumab IV over 1 hour on day 1. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Participants may continue on therapy beyond disease progression at the discretion of the investigator.
  Interventions: Biological: Durvalumab; Drug: Olaparib

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Drug: Olaparib — Given PO
  Other Names: AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281

SUMMARY:
This pilot phase I trial studies whether it is feasible to conduct a detailed molecular profile of triple negative breast cancer as part of a treatment strategy that asks whether or not we can lower the chance of breast cancer growing or spreading, by treating with a combination of PARP inhibitor how well (olaparib) and immune therapy (durvalumab). Olaparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving olaparib and durvalumab may work better in treating participants with metastatic triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the feasibility of completing Clinical Laboratory Improvement Act (CLIA) analytics on pre-treatment biopsy within a planned 4-week window for enrolled participants.

SECONDARY OBJECTIVES:

I. Assess safety and tolerability of the proposed therapy. II. Assess response to treatment. III. Determine the time to disease progression following study therapy. IV. Determine survival of participants enrolled on the study.

EXPLORATORY OBJECTIVES:

I. Examine response rates depending on tumor characteristics. II. Identify predictive biomarkers of sensitivity to therapy. III. Identify emerging mechanism of resistance to therapy tumor markers of emergence.

IV. Determine changes in tumor cells induced by PARP inhibitors. V. Identify tumor markers suggestive of combinatorial therapy that could r overcome resistance to therapy.

OUTLINE:

Participants receive olaparib orally (PO) twice a day (BID) for 28 days in the absence of disease progression or unacceptable toxicity. Participants then receive olaparib PO BID on days 1-28 and durvalumab intravenously (IV) over 1 hour on day 1. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Participants may continue on therapy beyond disease progression at the discretion of the investigator.

After completion of study treatment, participants are followed up every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Metastatic triple negative breast cancer (TNBC), as defined by:

  * Estrogen receptor (ER) and progesterone receptor (PR) negative as defined as ER < 10% and PR < 10% by immunohistochemistry according to American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines for hormone receptor testing
  * Human epidermal growth factor receptor 2 (HER2) non-amplified per ASCO/CAP guidelines, defined as:

    * immunohistochemistry (IHC) score 0/1+
    * IHC 2+ and in situ hybridization (ISH) non-amplified with a ratio of HER2 to CEP17 < 2.0, and if reported, average HER2 gene copy number < 4 signals/cells; or
    * ISH non-amplified with a ratio of HER2 to chromosome enumeration probe 17 (CEP17) < 2.0, and if reported, average HER2 gene copy number < 4 signals/cells
* Participants must have at least one measurable site of disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 that is amendable to biopsy.
* Prior therapies for metastatic breast cancer

  * Frontline patients who have not received prior systemic therapy for metastatic breast cancer are eligible,
  * Patients who have received =< 2 prior chemotherapy regimens for metastatic breast cancer are eligible
* Participants must have fully recovered from the acute toxic effects of all prior treatment to grade 1 or less, except alopecia and =< grade 2 neuropathy which are allowed
* Participants' life expectancy must be > 6 months
* Participant must have Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Participant must consent to undergo a pre-treatment screening biopsy for enrollment and subsequent biomarker analyses.
* Participants must consent to undergo one mandatory on-study tumor biopsy following a 4 week, single cycle induction treatment of olaparib. A second on-study biopsy at time of disease progression is optional, but not mandatory.
* Participants must not have had prior immunotherapy with anti-PD-L1, anti-PD-1, anti-CTLA4 or similar drugs.
* Participants must not have received previous treatment with PARP inhibitors
* Participants must not be planning to receive concomitantly other biologic therapy, hormonal therapy, other chemotherapy, surgery or other anti-cancer therapy except radiation therapy while receiving treatment on this protocol.
* Participant must be able to swallow tablets or capsules. A participant with any gastrointestinal disease that would impair ability to swallow, retain, or absorb drug is not eligible.
* Absolute neutrophil count (ANC) >= 1.5 x 10^9 /L (at time of registration and within 4 weeks prior to initiating on-protocol treatment)

  * May be waived on a case-by-case basis for patient populations recognized to have normal baseline values below this level.
* Platelets >= 100 x 10^9 /L (at time of registration and within 4 weeks prior to initiating on-protocol treatment)
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L (at time of registration and within 4 weeks prior to initiating on-protocol treatment)
* Creatinine =< 1.5 x upper limit of normal (ULN), OR measured or calculated creatinine clearance (glomerular filtration rate (GFR) can also be used in place of creatinine or CrCl) >= 60 mL/min/1.73m^2 for participants with creatinine levels > 1 x institutional ULN (at time of registration and within 4 weeks prior to initiating on-protocol treatment)

  * Creatinine clearance should be calculated per institutional standard. For participants with a baseline calculated creatinine clearance below normal institutional laboratory values, a measured baseline creatinine clearance should be determined. Individuals with higher values felt to be consistent with inborn errors of metabolism will be considered on a case-by-case basis.
* Total bilirubin =< 1.5 x ULN, OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN (at time of registration and within 4 weeks prior to initiating on-protocol treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN (at time of registration and within 4 weeks prior to initiating on-protocol treatment)
* Female participants of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female participants of childbearing potential must agree to use adequate methods of contraception starting with the first dose of study therapy through 60 days after the last dose of study therapy.

  * Participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year without an alternative medical cause.
  * Note: Abstinence is acceptable if this is the preferred contraception for the participant.
* Male participants must agree to use an adequate method of contraception starting with the first dose of study therapy through 60 days after the last dose of study therapy.

  * Note: Abstinence is acceptable if this is the preferred contraception for the participant.
* Participants must not have received live vaccines within 30 days prior to trial registration. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, shingles, yellow fever, rabies, bacillus Calmette-Guerin (BCG), and typhoid (oral) vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed.
* Participants must not have known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection prior to trial registration. Patients who have completed curative therapy for HCV are eligible. Patients with known human immunodeficiency virus (HIV) infection are eligible if they meet each of the following 3 criteria:

  * CD4 counts >= 350 mm^3
  * Serum HIV viral load of < 25,000 IU/ml and
  * Treated on a stable antiretroviral regimen.
* No other prior invasive malignancy is allowed except for the following: adequately treated basal (or squamous cell) skin cancer, in situ breast or cervical cancer. Stage I or II invasive cancer treated with a curative intent without evidence of disease recurrence for at least five years.

Exclusion Criteria:

* EXCLUSION - PARTICIPANT: Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 4 weeks of first dose of treatment.

  * Individuals in the follow-up phase of a prior investigational study may participate as long as it has been 4 weeks since last dose of the previous investigational agent of device.
* EXCLUSION - PARTICIPANT: Participant received prior chemotherapy or any other targeted therapies within the past 28, or palliative radiation within the past 14 days, prior to going on-study.
* EXCLUSION - PARTICIPANT: Participants with known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* EXCLUSION - PARTICIPANT: Participants with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging [confirmed by computed tomography (CT) scan if CT used at prior imaging, or confirmed by magnetic resonance imaging (MRI) if MRI was used at prior imaging) for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* EXCLUSION - PARTICIPANT: Active infection requiring systemic antibiotic therapy. Participants requiring systemic antibiotics for infection must have completed therapy before treatment is initiated.
* EXCLUSION - PARTICIPANT: Clinically significant cardiac disease or impaired cardiac function, including any of the following:

  * Clinically significant and/or uncontrolled heart disease such as congestive heart failure (New York Heart Association grade >= 2) uncontrolled hypertension, or clinically significant arrhythmia currently requiring medical treatment
  * Fridericia's correction formula (QTcF) > 470 msec for females, or > 450 msec for males, on screening electrocardiography (ECG) or congenital long QT syndrome
  * Acute myocardial infarction or unstable angina pectoris < 6 months prior to screening
* EXCLUSION - PARTICIPANT: Psychiatric illness/social situations that would limit compliance with study requirements
* EXCLUSION - PARTICIPANT: Participants with a history of hypersensitivity reactions to study agent or their excipients.
* EXCLUSION - PARTICIPANT: Participant is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* EXCLUSION - DURVALUMAB DRUG-SPECIFIC: Participant has evidence of interstitial lung disease or active non-infectious pneumonitis.
* EXCLUSION - DURVALUMAB DRUG-SPECIFIC: Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of durvalumab.

  * Note: Local surgery of isolated lesions for palliative intent is acceptable per investigator discretion.
* EXCLUSION - DURVALUMAB DRUG-SPECIFIC: Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* EXCLUSION - DURVALUMAB DRUG-SPECIFIC: Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

  * Participants with vitiligo or alopecia
  * Participants with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Participants without active disease in the last 5 years may be included but only after consultation with the study physician
  * Participants with celiac disease controlled by diet alone
* EXCLUSION - DURVALUMAB DRUG-SPECIFIC: History of allogenic organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Proportion of completion of Clinical Laboratory Improvement Act (CLIA) analytics on pre-treatment biopsy before the planned for 4-week biopsy | At day 28
  Using the feasibility analysis set, the proportion of the completed CLIA analytics within 4 weeks (i.e., from day 1, cycle 1 up to day 1 cycle 2 of on-study treatment regimen will be estimated relative to all screened participants who undergo a first biopsy with a 95% confidence interval.

SECONDARY OUTCOMES:
Incidence of >= grade 3 adverse events per Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.03 | Up to 3 months post treatment
  The incidence of having grade 3+ acute toxicity will be determined for participants with triple-negative breast cancer (TNBC) that received at least one dose of olaparib and durvalumab in combination. The 95% confidence interval will be reported with the point estimate of toxicity rate.
Overall response rate (ORR) for olaparib in combination with durvalumab | Up to 6 months post treatment
  The probability of having ORR will be measured and reported (if available) with 95% exact confidence interval.
Clinical benefit rate (CBR) for olaparib in combination with durvalumab | At 6 months post treatment
  CBR is defined as the percentage of participants who have achieved complete response, partial response and stable disease (i.e., CR + Pr + SD) at 6 months post-treatment. The probability of having CBR will be measured and reported (if available) with 95% exact confidence interval.
Duration of response (DOR) for olaparib in combination with durvalumab | Up to 6 months
  The duration of overall response is measured from the time measurement criteria are met for CR or Pr (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented taking as reference for progressive disease the smallest measurements recorded since the treatment started. The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that progressive disease is objectively documented. If a participant dies, irrespective of cause, without documentation of recurrent or progressive disease beforehand, then the date of death will be used to denote the response end date.
Progression-free survival (PFS) for olaparib in combination with durvalumab | Up to 1-year post treatment
  PFS is defined as the time from first treatment with olaparib (i.e., cycle 1 day 1) to the first of either recurrence or relapse (anywhere in the body), or death at time of last follow-up at 12-months. The estimated distribution of the PFS will be plotted using Kaplan Meier curves and reported with median survival and 95% confidence intervals if available.
Overall survival (OS) olaparib in combination with durvalumab | Up to 1-year post treatment
  OS is defined as the time from first treatment with olaparib (i.e., Day 1) to the date of death or last follow-up at 12 months. The estimated distribution of the OS will be plotted using Kaplan Meier curves and reported with median survival and 95% confidence intervals if available.

CONTACTS AND LOCATIONS:
Overall Officials: Zahi Mitri, MD, MS, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

REFERENCES:
- [Derived] Sun C, Fang Y, Labrie M, Li X, Mills GB. Systems approach to rational combination therapy: PARP inhibitors. Biochem Soc Trans. 2020 Jun 30;48(3):1101-1108. doi: 10.1042/BST20191092. PMID 32379297